CLINICAL TRIAL: NCT01230905
Title: Does Androgen Suppression Treatment In Prostate Cancer Reduce Myocardial Blood Flow Reserve?
Brief Title: Study to Monitor the Effects of Androgen Suppression Treatment on the Heart
Acronym: AST
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Responsible Party: Principal Investigator, Terrence Ruddy, Principal Investigator, Ottawa Heart Institute Research Corporation
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2008341-01H
Record Dates: First submitted 2010-10-28; First posted 2010-10-29 (Estimated); Last update posted 2017-04-24 (Actual); Status verified 2017-04

CONDITIONS: Prostate Cancer
Keywords: Androgen Suppression Therapy; Hormonal Toxicity; Quantitative PET; Myocardial blood flow; Coronary blood flow reserve; Endothelial dysfunction; Coronary Artery Disease
MeSH Terms: conditions — Prostatic Neoplasms; Coronary Artery Disease | interventions — Magnetic Resonance Spectroscopy; High-Energy Shock Waves

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MPI nuclear scan (Other): Nuclear MPI for CAD for prostate cancer subjects undergoing treatment and development of normal comparison.
  Interventions: Radiation: PET scan and ultrasound

INTERVENTIONS:
Radiation: PET scan and ultrasound — Nuclear rest/stress testing of the heart using N-13-ammonia paired with brachial artery ultrasound

SUMMARY:
Suppression of effects of androgens with male sex hormones, androgen suppression treatment (AST), has been known to reduce deaths and prolong life in advanced prostate cancer. There have, however, been concerns raised in previous studies that androgen suppression may be associated with increased rate of heart attacks, particularly in older men. This study looks at prostate cancer patients in The Ottawa Hospital Cancer Clinic to see if treating these patients with androgen suppression is associated with a decrease in blood flow to the heart muscles by using Positron Emission Tomography (PET) and brachial artery ultrasound.

DETAILED DESCRIPTION:
Treatment group: Prior to the initiation of AST, subjects will have a baseline N-13-ammonia PET scan and a brachial artery ultrasound at the University of Ottawa Heart Institute. Blood glucose and a lipid profile will be obtained. These tests will be repeated 6 - 9 months after starting AST.

Cancer control group: The same testing and intervals will be performed. Normals control group: Baseline testing will be done to establish a normal.

ELIGIBILITY:
Inclusion Criteria:

Cancer Population:

1. Diagnosis of prostate cancer
2. Treatment group: Scheduled to start AST, at Ottawa Hospital under the care of Radiation Oncology, Urology or Medical Oncology.

Control group: no AST scheduled as a treatment option for prostate cancer.

Non-Cancer Control Group

1. Male with low pre-test likelihood of coronary artery disease
2. No previous history of cancer.

Exclusion Criteria:

1. Known coronary disease including any of previous revascularization, history of myocardial infarction, coronary disease with >= 50% stenosis in a major coronary vessel on previous angiography, evidence of previous myocardial infarction on 12-lead electrocardiogram, positive myocardial perfusion scan, previous cardiac PET scan, stress echocardiogram or exercise stress test.
2. Subjects with a Summed Stress Score of >4 attributed to coronary disease on baseline PET images
3. Patients previously treated with AST
4. Patients with a life expectancy of less than 1 year.

Ages: 40 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 181 (Actual)
Dates: Start 2008-07; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
myocardial flow reserve | 6 - 9 months
  The change in global absolute MFR between baseline and follow up PET studies, at a patient level. MFR is defined as the ratio between regional blood flow with maximum vasodilation and baseline regional blood flow.

SECONDARY OUTCOMES:
Regional myocardial perfusion | 6 - 9 months
  The change in absolute MFR between baseline and follow up tests for the 3 major coronary territories. Territories with severe reduction in flow or no flow on baseline images will be censored from this analysis. Regional myocardial perfusion will be assessed semi-quantitatively by summed stress scores and summed difference scores in each of the PET scans in the treatment and control groups.
  Two-dimensional scans and pulse measures will be taken of the brachial artery with flow-mediated vasodilatation expressed as a percent change in arterial diameter from resting diameter.

CONTACTS AND LOCATIONS:
Overall Officials: Terrence Ruddy, MD, Principal Investigator — Ottawa Heart Institute Research Corporation
Locations (1):
- University of Ottawa Heart Institute, Ottawa, Ontario, Canada